CLINICAL TRIAL: NCT05273177
Title: Valutazione Della Funzione Neuromuscolare Dei Muscoli Flessori ed Estensori Del Ginocchio in Pazienti Con instabilità Cronica di Caviglia (CAI)
Brief Title: Muscle Strength Assessment in Patients With Chronic Ankle Instability
Acronym: KNEE-CAI
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Mariagrazia Benedetti, Professor, Istituto Ortopedico Rizzoli
Other Study IDs: PG. 0002018_2021
Record Dates: First submitted 2022-02-17; First posted 2022-03-10 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Chronic Ankle Instability
Keywords: ankle instability; muscle strength; quadriceps; hamstrings; maximal voluntary isometric contraction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAI group
  Interventions: Other: Chronic ankle instability
- Control group

INTERVENTIONS:
Other: Chronic ankle instability — Persistent condition of ankle instability after a first ankle sprain episode.
  Groups: CAI group

SUMMARY:
Patients with chronic ankle instability (CAI) show biomechanical and neuromuscular alterations during the performance of functional movements not only at the ankle joint level, but also in more proximal joints and segments. Few studies have been conducted to investigate the effects of chronic ankle instability on neuromuscular control at the knee joint level. The aim of this study is to investigate whenther abnormalities exists in maximal and sub-maximal isometric muscle strength expression in patients with CAI.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 40 years
* chronic ankle instability
* physically active individuals

Exclusion Criteria:

* sedentary behaviour
* previous injuries or surgeries to the lower limbs
* neurological disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Orthopaedic hospital and community individuals
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Forces exerted by knee extensor and flexor muscles | Day 1
  The forces (N) exerted by knee extensor and flexor muscles will be assessed by means of a dynamometer during maximal and submaximal isometric muscle contractions.

SECONDARY OUTCOMES:
Knee extensor and flexor muscles activations | Day 1
  Knee extensor and flexor muscles activations (mV) during the maximal and submaximal isometric contractions will be recorded by means of surface electrodes for electromyography.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Benedetti, MD, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Labanca L, Tedeschi R, Mosca M, Benedetti MG. Individuals With Chronic Ankle Instability Show Abnormalities in Maximal and Submaximal Isometric Strength of the Knee Extensor and Flexor Muscles. Am J Sports Med. 2024 Apr;52(5):1328-1335. doi: 10.1177/03635465241232090. Epub 2024 Mar 8. PMID 38459686